CLINICAL TRIAL: NCT02345486
Title: Isotonic Solution Administration Logistical Testing: Pilot Study for the Isotonic Solutions and Major Adverse Renal Events Trial
Brief Title: Isotonic Solution Administration Logistical Testing
Acronym: SALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Todd Rice, Assistant Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 141349
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Acute Kidney Injury
Keywords: Pilot Projects; Plasmalyte A; Ringer's lactate; Sodium Chloride; Critical Care; Resuscitation"
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Chloride; Ringer's Lactate; Plasmalyte A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.9% sodium chloride (Active Comparator): Participants in the '0.9% sodium chloride' arm will receive 0.9% sodium chloride ('normal saline') any time an isotonic crystalloid is ordered by a provider during the intensive care unit admission.
  Interventions: Other: 0.9% sodium chloride
- Physiologically balanced fluid (Active Comparator): Participants in the 'physiologically balanced fluid' arm will receive physiologically balanced fluid (Lactated ringers or Plasmalyte-A) any time an isotonic crystalloid is ordered by a provider during the intensive care unit admission.
  Interventions: Other: Physiologically balanced fluid

INTERVENTIONS:
Other: 0.9% sodium chloride
  Arms: 0.9% sodium chloride
Other: Physiologically balanced fluid
  Other Names: Lactated ringers or Plasmalyte-A
  Arms: Physiologically balanced fluid

SUMMARY:
The administration of intravenous crystalloids is ubiquitous in the care of the critically ill. Commonly available crystalloid solutions contain a broad spectrum of electrolyte compositions including a range of chloride concentrations. Recent studies of associated higher fluid chloride content with acute kidney injury and mortality but no large, randomized trials have been conducted. In preparation for a large, cluster-randomized, multiple-crossover trial comparing 0.9% sodium chloride to physiologically-balanced isotonic crystalloids (Lactated Ringers or Plasmalyte-A) in intensive care unit patients, this pilot study will enroll all patients admitted to the medical intensive care unit at a single tertiary center for a sixth month period. The primary objective will be to test the ability of an electronic order entry tool to ensure administration of assigned study fluid or record contraindications to assigned study fluid. The pilot study will also demonstrate the feasibility of collecting demographic, severity of illness, fluid management, vital sign, laboratory, acute kidney injury and renal replacement therapy, and outcome data in an automated, electronic fashion.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the adult medical intensive care unit (MICU) at Vanderbilt University Medical Center

Exclusion Criteria:

* Age<18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd W Rice, M.D., M.Sc., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Yunos NM, Kim IB, Bellomo R, Bailey M, Ho L, Story D, Gutteridge GA, Hart GK. The biochemical effects of restricting chloride-rich fluids in intensive care. Crit Care Med. 2011 Nov;39(11):2419-24. doi: 10.1097/CCM.0b013e31822571e5. PMID 21705897
- [Background] Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. JAMA. 2012 Oct 17;308(15):1566-72. doi: 10.1001/jama.2012.13356. PMID 23073953
- [Background] Raghunathan K, Shaw A, Nathanson B, Sturmer T, Brookhart A, Stefan MS, Setoguchi S, Beadles C, Lindenauer PK. Association between the choice of IV crystalloid and in-hospital mortality among critically ill adults with sepsis*. Crit Care Med. 2014 Jul;42(7):1585-91. doi: 10.1097/CCM.0000000000000305. PMID 24674927
- [Derived] Semler MW, Wanderer JP, Ehrenfeld JM, Stollings JL, Self WH, Siew ED, Wang L, Byrne DW, Shaw AD, Bernard GR, Rice TW; SALT Investigators * and the Pragmatic Critical Care Research Group; SALT Investigators. Balanced Crystalloids versus Saline in the Intensive Care Unit. The SALT Randomized Trial. Am J Respir Crit Care Med. 2017 May 15;195(10):1362-1372. doi: 10.1164/rccm.201607-1345OC. PMID 27749094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This cluster-randomized, multiple-crossover trial enrolled 974 adults admitted to a tertiary medical intensive care unit from February 3, 2015 to May 31, 2015.
Groups:
- 0.9% Sodium Chloride: Participants in the '0.9% sodium chloride' arm will receive 0.9% sodium chloride ('normal saline') any time an isotonic crystalloid is ordered by a provider during the intensive care unit admission.
  0.9% sodium chloride
- Physiologically Balanced Fluid: Participants in the 'physiologically balanced fluid' arm will receive physiologically balanced fluid (Lactated ringers or Plasmalyte-A) any time an isotonic crystalloid is ordered by a provider during the intensive care unit admission.
  Physiologically balanced fluid
Period: Overall Study
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Started | 454 | 520
Completed | 454 | 520
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid | Total
Number analyzed (Participants) | 454 | 520 | 974
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [46 to 70] | 57 [44 to 68] | 58 [45 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 252 | 460
  Male | 246 | 268 | 514
Region of Enrollment [Number; unit: participants]
  United States | 454 | 520 | 974
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] — Body mass index, median (IQR), kg/m2
  kg/m^2 | 26.4 [22.4 to 32.8] | 26.7 [22.5 to 32.5] | 26.6 [22.5 to 32.7]
Chronic kidney disease, stage III or greater [Count of Participants; unit: Participants] | 104 | 119 | 223
Previous renal replacement therapy [Count of Participants; unit: Participants] | 44 | 42 | 86
Source of ICU Admission [Count of Participants; unit: Participants]
  Emergency Department | 256 | 310 | 566
  Transfer from another hospital | 93 | 106 | 199
  Hospital ward | 80 | 79 | 159
  Another ICU within the hospital | 15 | 14 | 29
  Operating room | 6 | 4 | 10
  Outpatient | 4 | 7 | 11
Mechanical ventilation [Count of Participants; unit: Participants] | 155 | 174 | 329
Vasopressors [Count of Participants; unit: Participants] | 111 | 114 | 225
Acute kidney injury, stage II or greater [Count of Participants; unit: Participants] | 87 | 96 | 183

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Isotonic Crystalloid Which is 0.9% Saline
Description: Proportion of total intravenous isotonic crystalloid administered during admission to the intensive care unit that is 0.9% sodium chloride, censored at 30 days. The primary outcome was the proportion of intravenous isotonic crystalloid administered in the ICU that was saline. This was a continuous variable calculated for each patient as the volume of saline received divided by volume of saline received plus volume of balanced crystalloids received with a range from 0.0 (no saline received) to 1.0 (only saline received).
Time Frame: 30 days
Measure: Mean (Full Range); unit: Percentage of fluid that was saline
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Percentage of fluid that was saline | 91.2 [0 to 100] | 21.0 [0 to 100]
Statistical Analysis 1: Comparison: 0.9% Sodium Chloride vs Physiologically Balanced Fluid; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.70, 95% CI 2-sided [0.66 to 0.74] — reported "mean difference" is a difference in proportions

2. Secondary Outcome: Proportion of Isotonic Crystalloid Which is Physiologically Balanced
Description: Proportion of total intravenous isotonic crystalloid administered during admission to the intensive care unit that is either Lactated ringers or Plasmalyte-A, censored at 30 days.
Time Frame: 30 days
Measure: Mean (Full Range); unit: Percentage of fluid that was balanced
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Percentage of fluid that was balanced | 8.8 [0 to 100] | 78.8 [0 to 100]

3. Secondary Outcome: Total Intravenous Input
Description: Total volume of intravenous fluid administration during admission to the intensive care unit, censored at 30 days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
milliliters | 2000 [792 to 4630] | 2125 [1000 to 4625]

4. Secondary Outcome: Total Isotonic Crystalloid Input
Description: Total volume of intravenous isotonic crystalloid administration during admission to the intensive care unit, censored at 30 days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
mL | 1424 [500 to 3377] | 1617 [500 to 3628]

5. Secondary Outcome: Total Intravenous Colloid Input
Description: Total volume of intravenous colloid administration (excluding blood products) during admission to the intensive care unit, censored at 30 days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
milliliters | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Total Intravenous Blood Product Administration
Description: Total volume of packed red blood cells, platelets, and fresh frozen plasma administered during admission to the intensive care unit, censored at 30 days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
milliliters | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Highest Serum Chloride Between Enrollment and Day 30
Description: highest serum chloride (mmol/L) during admission to the intensive care unit, censored at 30 days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
mmol/L | 109 [105 to 113] | 108 [104 to 112]

8. Secondary Outcome: Highest Serum Sodium Between Enrollment and Day 30
Description: Highest serum sodium concentration (mmol/L) during admission to the intensive care unit, censored at 30 days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
mmol/L | 141 [139 to 144] | 141 [138 to 144]

9. Secondary Outcome: Lowest Bicarbonate Concentration Between Enrollment and Day 30
Description: Lowest serum bicarbonate concentration (mmol/L) during admission to the intensive care unit, censored at 30 days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
mmol/L | 19 [16 to 22] | 19 [15 to 22]

10. Secondary Outcome: Number of Patients With MAKE30
Description: Incidence of Major Adverse Kidney Events by 30 days -- a composite outcome defined as one or more of the following: death, new use of renal replacement therapy, or persistence of renal dysfunction at hospital discharge or at 30 days (defined as an increase in serum creatinine ≥ 200% from baseline)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Participants | 112 | 128

11. Secondary Outcome: In-hospital Mortality
Description: Death prior to the earlier of hospital discharge or day 30
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Participants | 68 | 72

12. Secondary Outcome: New Use of Renal Replacement Therapy
Description: Receipt of new renal replacement therapy after the first study day, censored at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Participants | 14 | 24

13. Secondary Outcome: Persistent Renal Dysfunction
Description: Persistence of renal dysfunction at hospital discharge or at 30 days (defined as an increase in serum creatinine ≥ 200% from baseline)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Participants | 59 | 76

14. Secondary Outcome: Number of Contraindications
Description: Number of contraindications to assigned study fluid identified by providers, censored at 30 days
Time Frame: 30 days
Population: Order for intravenous crystalloid is the unit analyzed; each patient could have multiple orders for intravenous crystalloid
Measure: Count of Units; unit: Orders for intravenous crystalloid
Units Other Than Participants: Orders for intravenous crystalloid
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Number analyzed (Orders for intravenous crystalloid) | 588 | 854
Orders for intravenous crystalloid | 28 | 66

15. Secondary Outcome: Incidence of Hyperchloremia
Description: Incidence of hyperchloremia defined as a serum chloride greater than or equal to 110 mmol/L
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Participants | 171 | 171

16. Secondary Outcome: Incidence of Severe Hypochloremia
Description: Incidence of severe hypochloremia defined as a serum chloride less than 90mmol/L
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Participants | 34 | 32

17. Secondary Outcome: Increase in Serum Creatinine
Description: Increase in serum creatinine during hospitalization, censored at 30 days Change from baseline to highest value, median (IQR), mg/dl
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
mg/dL | 0.07 [-0.1 to 0.5] | 0.07 [-0.1 to 0.5]

18. Secondary Outcome: Incidence of Acute Kidney Injury
Description: Incidence of stage II or III acute kidney injury by Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury criteria, censored at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
Participants | 129 | 135

19. Secondary Outcome: Intensive Care Unit Free Days to Day 28
Description: ICU-free days to 28 days after enrollment will be defined as the number of days alive and not admitted to an intensive care unit service after the patient's final discharge from the intensive care unit before 28 days. If the patient is admitted to an intensive care unit service at day 28 or dies prior to day 28, ICU-free days will be 0.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
days | 25.1 [22.1 to 26.2] | 25.2 [21.8 to 26.4]

20. Secondary Outcome: Ventilator-free Days (VFD) to Day 28
Description: Ventilator-free days to day 28 will be defined as the number of days alive and with unassisted breathing to day 28 after enrollment, assuming a patient survives for at least two consecutive calendar days after initiating unassisted breathing and remains free of assisted breathing. If a patient returns to assisted breathing and subsequently achieves unassisted breathing prior to day 28, VFD will be counted from the end of the last period of assisted breathing to day 28. If the patient is receiving assisted ventilation at day 28 or dies prior to day 28, VFD will be 0.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
days | 28.0 [27.0 to 28.0] | 28.0 [26.0 to 28.0]

21. Secondary Outcome: Dialysis-free Survival to Day 28
Description: Dialysis free survival to day 28 will be defined as the number of days alive and without dialysis receipt to day 28 after enrollment, assuming a patient survives for at least two consecutive calendar days after last receipt of dialysis and remains free of dialysis. If the patient is receiving dialysis at day 28 or dies prior to day 28, VFD will be 0.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
days | 28.0 [28.0 to 28.0] | 28.0 [28.0 to 28.0]

22. Secondary Outcome: Peak Creatinine in the First 30 Days
Description: Highest creatinine value in the first 30 days
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
Number analyzed (Participants) | 454 | 520
mg/dL | 1.19 [0.81 to 2.30] | 1.19 [0.80 to 2.62]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 0.9% Sodium Chloride | Physiologically Balanced Fluid
All-Cause Mortality (participants affected / at risk) | 68/454 | 72/520
Serious Adverse Events (participants affected / at risk) | 0/454 | 0/520
Other Adverse Events (participants affected / at risk) | 0/454 | 0/520

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes